CLINICAL TRIAL: NCT02978573
Title: A Post Approval Study to Evaluate the Safety and Effectiveness of Cartiva Implant in the Treatment of First Metatarsophalangeal Joint Osteoarthritis as Compared to a Control
Brief Title: Post Approval Study to Evaluate the Effectiveness and Safety of Cartiva Implant in the Treatment of OA of the Great Toe
Acronym: MOTION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cartiva, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC-0031 (PAS)
Record Dates: First submitted 2016-11-11; First posted 2016-12-01 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis of First Metatarsalphalangeal Joint
Keywords: First MTP Joint; Hallux Rigidus; Hallux Limitus; Cartilage Replacement; Osteoarthritis; First MTP Joint Osteoarthritis; Big Toe Pain
MeSH Terms: conditions — Hallux Rigidus; Hallux Limitus; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cartiva (Experimental): Cartiva Synthetic Cartilage Implant
  Interventions: Device: Cartiva

INTERVENTIONS:
Device: Cartiva — Cartiva Synthetic Cartilage Implant

SUMMARY:
Evaluate and confirm the long-term safety and effectiveness of the Cartiva SCI implant established by the pivotal trial.

DETAILED DESCRIPTION:
As part of the Conditions of Approval of Cartiva SCI for the treatment of first MTP osteoarthritis, the Food and Drug Administration (FDA) requires additional long term data to evaluate the long term safety and effectiveness of Cartiva including the durability and survivorship of the implant. This Post-Approval Study (PAS) addendum is intended to supplement the initial 24 months follow up period and provide additional long term safety and effectiveness data on Cartiva

ELIGIBILITY:
Inclusion Criteria:

* Subject must have been treated with Cartiva under MOTION study protocol PTC-0031; and,
* Have been informed of the nature of the study, agreeing to its requirements, and have signed the informed consent approved by the IRB/Ethics Committee for long-term follow-up.

Exclusion Criteria:

* Subjects who underwent a secondary surgical intervention to have the Cartiva implant removed during the 24-month time period of participation in the MOTION study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
Long Term Safety of the Cartiva Implant by demonstrating durability over the long term and no unanticipated safety concerns that arise | 5 year
  1. Durability of the implant over the longer term. This will be addressed using survival analysis starting at Month 24 to determine the rate of implant removals among devices that survived to Month 24. A complementary survival analysis starting at index surgery to end of study will also be performed.
  2. There are no unanticipated safety concerns that arise after Month 24 up to 5 years. This will be addressed by a) determining the incidence of serious device-related adverse events per year and overall from Month 24 to Year 5; and b) summarizing device-related radiographic complications1 over time from Month 24 to Year 5. Note that this analysis will address both device and procedure related complications and serious device-related adverse events whether observed previously in the 24 month follow up portion of the study or encountered for this first time during the extended follow-up period.

SECONDARY OUTCOMES:
Pain Scale (VAS) | 5 year
  Visual Analog Scale (VAS) Pain
Foot and Ankle Ability Measure (FAAM) Activities of Daily Living (ADL) | 5 year
  Foot and Ankle Ability Measure (FAAM) Activities of Daily Living scores
Foot and Ankle Ability Measure (FAAM) Sports | 5 year
  Foot and Ankle Ability Measure (FAAM) Sports scores

CONTACTS AND LOCATIONS:
Overall Officials: Judith Baumhauer, MD, Principal Investigator — University of Rochester

IPD SHARING:
Plan to Share IPD: No